CLINICAL TRIAL: NCT01243762
Title: Phase I Parallel Arm Study of MK-0646 (Dalotuzumab) + MK-2206, Dalotuzumab + MK-0752, and Dalotuzumab + MK-8669 (Ridaforolimus) Doublets (MK-MK Doublets) in Patients With Advanced Cancer
Brief Title: A Study of Dalotuzumab + MK-2206, Dalotuzumab + MK-0752, and Dalotuzumab + Ridaforolimus Combination Therapies in Participants With Advanced Cancer (MK-0646-027)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated for business reasons and not due to any safety or efficacy concerns related to dalotuzumab.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0646-027
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2017-10-30 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Neoplasms Malignant
Keywords: Colorectal cancer; Solid tumors; Ovarian cancer; Fallopian tube cancer; Primary peritoneal cancer
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — dalotuzumab; 3-(4-((4-chlorophenyl)sulfonyl)-4-(2,5-difluorophenyl)cyclohexyl)propanoic acid; ridaforolimus; MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg (Experimental): Participants in Part 1 of the study receive dalotuzumab 7.5 mg/kg intravenously (IV) weekly + MK-0752 1800 mg orally (PO) weekly in 28-day cycles for a maximum of 6 months of study therapy.
  Interventions: Drug: dalotuzumab; Drug: MK-0752
- Dalotuzumab 10 mg/kg + MK-0752 1800 mg (Experimental): Participants in Parts 1 and 2 of the study receive dalotuzumab 10 mg/kg IV weekly + MK-0752 1800 mg PO weekly in 28-day cycles for a maximum of 6 months of study therapy.
  Interventions: Drug: dalotuzumab; Drug: MK-0752
- Dalotuzumab 10 mg/kg + MK-2206 90 mg (Experimental): Participants in Part 1 of the study receive dalotuzumab 10 mg/kg IV weekly + MK-2206 90 mg PO weekly in 28-day cycles for a maximum of 6 months of study therapy.
  Interventions: Drug: dalotuzumab; Drug: MK-2206
- Dalotuzumab 10 mg/kg + MK-2206 135 mg (Experimental): Participants in Part 1 of the study receive dalotuzumab 10 mg/kg IV weekly + MK- 2206 135 mg PO weekly in 28-day cycles for a maximum of 6 months of study therapy.
  Interventions: Drug: dalotuzumab; Drug: MK-2206
- Dalotuzumab 10 mg/kg + MK-2206 150 mg (Experimental): Participants in Parts 1 and 2 of the study receive dalotuzumab 10 mg/kg IV weekly + MK- 2206 150 mg PO weekly in 28-day cycles for a maximum of 6 months of study therapy.
  Interventions: Drug: dalotuzumab; Drug: MK-2206
- Dalotuzumab 10 mg/kg + MK-2206 200 mg (Experimental): Participants in Part 1 of the study receive dalotuzumab 10 mg/kg IV weekly + MK- 2206 200 mg PO weekly in 28-day cycles for a maximum of 6 months of study therapy.
  Interventions: Drug: dalotuzumab; Drug: MK-2206
- Dalotuzumab + Ridaforolimus (Experimental): Participants in Part 2 of the study receive dalotuzumab 10 mg/kg IV weekly + ridaforolimus 20 mg PO daily for 5 consecutive days per week in 28-day cycles for a maximum of 6 months of study therapy.
  Interventions: Drug: dalotuzumab; Drug: ridaforolimus

INTERVENTIONS:
Drug: dalotuzumab — Administered intravenously (IV) once weekly in 28-day cycles for a maximum of 6 months of study therapy
  Other Names: MK-0646
Drug: MK-0752 — Administered orally (PO) weekly in 28-day cycles for a maximum of 6 months of study therapy
  Arms: Dalotuzumab 10 mg/kg + MK-0752 1800 mg; Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg
Drug: ridaforolimus — Administered PO daily for 5 consecutive days per week in 28-day cycles for a maximum of 6 months of study therapy
  Other Names: MK-8669
  Arms: Dalotuzumab + Ridaforolimus
Drug: MK-2206 — Administered PO weekly in 28-day cycles for a maximum of 6 months of study therapy
  Arms: Dalotuzumab 10 mg/kg + MK-2206 135 mg; Dalotuzumab 10 mg/kg + MK-2206 150 mg; Dalotuzumab 10 mg/kg + MK-2206 200 mg; Dalotuzumab 10 mg/kg + MK-2206 90 mg

SUMMARY:
This is an open-label, two-part study to evaluate the safety and tolerability of combination treatment with dalotuzumab + MK-2206, dalotuzumab + MK-0752, or dalotuzumab + ridaforolimus (MK-8669). Part 1 of the study will determine the dose-limiting toxicities (DLTs) observed after administration of each of the combinations at various doses and define the maximum tolerated dose (MTD) of each combination. Part 2 of the study will assess preliminary anti-tumor activity of these combinations (at MTD) in two groups of participants with selected tumor biomarkers: one group with metastatic or recurrent platinum-resistant ovarian cancer, fallopian tube cancer, or primary peritoneal cancer and one group with metastatic or recurrent colorectal cancer. The dalotuzumab + ridaforolimus and dalotuzumab + MK-2206 arms will be enriched with female platinum-resistant ovarian cancer, fallopian tube cancer, or primary peritoneal cancer participants. The dalotuzumab + MK-0752 arm will be enriched with metastatic or recurrent wild-type kirsten rat sarcoma (KRAS) colorectal cancer participants.

The primary hypothesis is that the DLTs observed in adult patients with locally advanced or metastatic solid tumors after administration of each of the MK-MK doublets will be dose-dependent to allow for definition of a MTD within each MK-MK doublet.

ELIGIBILITY:
Inclusion Criteria:

* Participants must not have any medical conditions that may impact compliance with the protocol, limit interpretation of study results, or pose an unacceptable medical risk.
* Participant must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (EGOG) Performance Scale.
* Participant is able to swallow capsules and has no condition that will preclude swallowing and absorbing oral medications on an ongoing basis.
* Participant has no history of a prior malignancy with the exception of cervical intraepithelial neoplasia; basal cell carcinoma of the skin; adequately treated localized prostate carcinoma with prostatic specific antigen (PSA) < 1.0; or has undergone potentially curative therapy with no evidence of that disease for five years, or is deemed at low risk for recurrence by his/her treating physician.
* Participant has at least one measurable metastatic or recurrent lesion according to Response Criteria in Solid Tumors (RECIST).

Part 1:

* Participant must have a histologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist, or participant is not a candidate for standard therapy, or is unwilling to undergo standard therapy. There is no limit on the number of prior treatment regimens.

Part 2:

* A female participant assigned to the dalotuzumab + MK-2206 or dalotuzumab + ridaforolimus treatment arms must have histologically-confirmed metastatic or recurrent platinum-resistant ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist, or participant is not a candidate for standard therapy, or is unwilling to undergo standard therapy. Participants may have received any number of prior treatment regimens.
* A participant assigned to the dalotuzumab + MK-0752 treatment arms must have histologically-confirmed metastatic or recurrent wild-type KRAS colorectal cancer that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist, or participant is not a candidate for standard therapy, or is unwilling to undergo standard therapy. Participants may have received any number of prior treatment regimens.
* Participant agrees to provide archival tumor tissue sample or undergo biopsy for analysis of gene expression levels.

Exclusion Criteria:

* Participant has had chemotherapy, radiotherapy, or biological therapy (including monoclonal antibodies) within 4 weeks prior to study Day 1 (6 weeks for nitrosoureas or mitomycin C) or who has not recovered from adverse events due to agents administered more than 4 weeks earlier, or major surgery <4 weeks earlier.
* Participant is currently participating or has participated in a study with an investigational compound or device within 28 days, or 5X half-life of the investigational compound (excluding monoclonal antibodies), whichever is longer, of initial dosing on this study. Participants previously treated with a monoclonal antibody will be eligible to participate after a 28 day washout period.
* Participants with known central nervous system (CNS) metastases and/or carcinomatous meningitis are excluded.
* Participant has significant or uncontrolled cardiovascular disease, including New York Heart Association (NYHA) Class III-IV heart failure, unstable angina, or a myocardial infarction within the last 6 months.
* Participant is known to have diabetes that is poorly controlled.
* Participant is pregnant, breastfeeding, or expecting to conceive or father children during the study.
* Participant is known to be human immunodeficiency virus (HIV)-positive.
* Participant has active Hepatitis B or C infection.
* Participant has symptomatic ascites or pleural effusion.
* Participant requires treatment with immunosuppressive agents other than prescribed corticosteroids at stable doses for at least two weeks prior to the first dose of study drug.
* Participant requires treatment with medication(s) that strongly or moderately induce or inhibit cytochrome P450.
* Participant is using growth hormone or growth hormone inhibitors.
* Participant requires treatment with therapeutic warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2012-12-04 (Actual); Study Completion 2013-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Brana I, Berger R, Golan T, Haluska P, Edenfield J, Fiorica J, Stephenson J, Martin LP, Westin S, Hanjani P, Jones MB, Almhanna K, Wenham RM, Sullivan DM, Dalton WS, Gunchenko A, Cheng JD, Siu LL, Gray JE. A parallel-arm phase I trial of the humanised anti-IGF-1R antibody dalotuzumab in combination with the AKT inhibitor MK-2206, the mTOR inhibitor ridaforolimus, or the NOTCH inhibitor MK-0752, in patients with advanced solid tumours. Br J Cancer. 2014 Nov 11;111(10):1932-44. doi: 10.1038/bjc.2014.497. Epub 2014 Oct 7. PMID 25290091

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 participants enrolled in Part 1 (dose escalation/preliminary maximum tolerated dose [MTD] identification). 12 participants continued in Part 2 (preliminary anti-tumor activity assessment), and 6 new participants were enrolled in Part 2 that did not participate in Part 1 (total enrollment = 47). Study terminated prior to completion of Part 2.
Groups:
- Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg: Participants received dalotuzumab 7.5 mg/kg IV weekly + MK-0752 1800 mg PO weekly in 28-day cycles for a minimum of 6 cycles until disease progression or study discontinuation.
- Dalotuzumab 10 mg/kg + MK-0752 1800 mg: Participants received dalotuzumab 10 mg/kg IV weekly + MK-0752 1800 mg PO weekly in 28-day cycles for a minimum of 6 cycles until disease progression or study discontinuation.
- Dalotuzumab 10 mg/kg + MK-2206 90 mg: Participants received dalotuzumab 10 mg/kg IV weekly + MK-2206 90 mg PO weekly in 28-day cycles for a minimum of 6 cycles until disease progression or study discontinuation.
- Dalotuzumab 10 mg/kg + MK-2206 135 mg: Participants received dalotuzumab 10 mg/kg IV weekly + MK-2206 135 mg PO weekly in 28-day cycles for a minimum of 6 cycles until disease progression or study discontinuation.
- Dalotuzumab 10 mg/kg + MK-2206 150 mg: Participants received dalotuzumab 10 mg/kg IV weekly + MK-2206 150 mg PO weekly in 28-day cycles for a minimum of 6 cycles until disease progression or study discontinuation.
- Dalotuzumab 10 mg/kg + MK-2206 200 mg: Participants received dalotuzumab 10 mg/kg IV weekly + MK-2206 200 mg PO weekly in 28-day cycles for a minimum of 6 cycles until disease progression or study discontinuation.
- Dalotuzumab + Ridaforolimus: Participants received dalotuzumab 10 mg/kg IV weekly + ridaforolimus 20 mg PO daily for 5 consecutive days per week in 28-day cycles for a minimum of 6 cycles until disease progression or study discontinuation.
Period: Part 1 (Dose Escalation/MTD)
Arm/Group | Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-2206 90 mg | Dalotuzumab 10 mg/kg + MK-2206 135 mg | Dalotuzumab 10 mg/kg + MK-2206 150 mg | Dalotuzumab 10 mg/kg + MK-2206 200 mg | Dalotuzumab + Ridaforolimus
Started | 4 | 13 | 3 | 8 | 10 | 3 | 0
Completed | 1 (Entered Part 2 of Study) | 5 (Entered Part 2 of Study) | 0 | 2 (Entered Part 2 of Study) | 4 (Entered Part 2 of Study) | 0 | 0
Not Completed | 3 | 8 | 3 | 6 | 6 | 3 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 2 | 3 | 5 | 5 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Dose Confirmation/Efficacy)
Arm/Group | Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-2206 90 mg | Dalotuzumab 10 mg/kg + MK-2206 135 mg | Dalotuzumab 10 mg/kg + MK-2206 150 mg | Dalotuzumab 10 mg/kg + MK-2206 200 mg | Dalotuzumab + Ridaforolimus
Started | 1 | 5 | 0 | 2 | 4 | 0 | 6 (New participants were enrolled in Part 2 of the study that did not participate in Part 1)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 5 | 0 | 2 | 4 | 0 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 3
Not completed — Progressive Disease | 1 | 3 | 0 | 1 | 2 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number of participants for each dose combination for the overall study
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-2206 90 mg | Dalotuzumab 10 mg/kg + MK-2206 135 mg | Dalotuzumab 10 mg/kg + MK-2206 150 mg | Dalotuzumab 10 mg/kg + MK-2206 200 mg | Dalotuzumab + Ridaforolimus | Total
Number analyzed (Participants) | 4 | 13 | 3 | 8 | 10 | 3 | 6 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (4.6) | 59.0 (12.2) | 50.3 (12.7) | 60.4 (12.0) | 65.4 (7.0) | 57.3 (10.1) | 68.8 (14.1) | 60.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 2 | 4 | 4 | 3 | 6 | 33
  Male | 1 | 2 | 1 | 4 | 6 | 0 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as follows: 1) non-hematological toxicity ≥Grade 3 according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 except for Grade 3 nausea, vomiting, diarrhea, and/or dehydration; Grade 3 or 4 hyperglycemia; alopecia; inadequately treated hypersensitivity reactions; dalotuzumab infusion-related reactions; Grade 3 transaminases ≤1 week in duration; or clinically non-significant, treatable or reversible lab abnormalities; 2) Grade 4-5 hematologic toxicity, with the exception of Grade 4 neutropenia <6 days in duration; 3) Grade 3 or Grade 4 neutropenia with fever >38.5 degrees C; 4) Grade 4 thrombocytopenia ≤25.0 x 10^9/Liter; 5) drug-related adverse experience leading to a dose modification during Cycle 1; 6) unresolved drug-related toxicity that causes ≥3 week delay of the next scheduled dose of study medication; 7) persistent increases in QTc interval >60 milliseconds from baseline, or clinically significant bradycardia.
Time Frame: Cycle 1-28 Days
Population: All participants who completed the first cycle of study therapy or discontinued from the study due to a DLT attributable to study therapy.
Measure: Number; unit: Participants
Arm/Group | Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-2206 90 mg | Dalotuzumab 10 mg/kg + MK-2206 135 mg | Dalotuzumab 10 mg/kg + MK-2206 150 mg | Dalotuzumab 10 mg/kg + MK-2206 200 mg | Dalotuzumab + Ridaforolimus
Number analyzed (Participants) | 4 | 13 | 3 | 8 | 10 | 3 | 3
Participants | 1 | 3 | 0 | 1 | 3 | 2 | 0

2. Secondary Outcome: Number of Participants Whose Best Response is a Partial Response (PR) or Complete Response (CR)
Description: Best response was determined for the maximum tolerated dose from the start of treatment until disease progression, recurrence, or completion of 6 months of treatment. Lesions were measured by computed tomography (CT) scan or magnetic resonance imaging (MRI). Partial response (PR), defined as a tumor burden decrease of 30%, or complete response (CR) was determined using Response Criteria in Solid Tumors (RECIST) 1.1 for participants with at least one measurable target lesion at baseline.
Time Frame: Up to 7 months
Population: All participants who received at least one dose of study therapy and had baseline data for those analyses that required baseline data. The analysis was planned to be performed on the 3 arms in Part 2 only. The study was terminated prior to completion of this analysis.
Measure: Number; unit: Participants
Arm/Group | Dalotuzumab 10 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-2206 150 mg | Dalotuzumab + Ridaforolimus
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: Adverse events collected for all participants who received at least one dose of study therapy
Arm/Group | Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-0752 1800 mg | Dalotuzumab 10 mg/kg + MK-2206 90 mg | Dalotuzumab 10 mg/kg + MK-2206 135 mg | Dalotuzumab 10 mg/kg + MK-2206 150 mg | Dalotuzumab 10 mg/kg + MK-2206 200 mg | Dalotuzumab + Ridaforolimus
Serious Adverse Events (participants affected / at risk) | 2/4 | 6/13 | 0/3 | 3/8 | 6/10 | 3/3 | 5/6
Other Adverse Events (participants affected / at risk) | 4/4 | 13/13 | 3/3 | 8/8 | 10/10 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg (N=4) | Dalotuzumab 10 mg/kg + MK-0752 1800 mg (N=13) | Dalotuzumab 10 mg/kg + MK-2206 90 mg (N=3) | Dalotuzumab 10 mg/kg + MK-2206 135 mg (N=8) | Dalotuzumab 10 mg/kg + MK-2206 150 mg (N=10) | Dalotuzumab 10 mg/kg + MK-2206 200 mg (N=3) | Dalotuzumab + Ridaforolimus (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 7.5 mg/kg + MK-0752 1800 mg (N=4) | Dalotuzumab 10 mg/kg + MK-0752 1800 mg (N=13) | Dalotuzumab 10 mg/kg + MK-2206 90 mg (N=3) | Dalotuzumab 10 mg/kg + MK-2206 135 mg (N=8) | Dalotuzumab 10 mg/kg + MK-2206 150 mg (N=10) | Dalotuzumab 10 mg/kg + MK-2206 200 mg (N=3) | Dalotuzumab + Ridaforolimus (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Orbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (2) | 4 (4) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 5 (7) | 1 (1) | 4 (5) | 4 (4) | 1 (1) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 10 (10) | 1 (2) | 4 (5) | 3 (3) | 2 (4) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (4) | 7 (7) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (4)
Asthenia (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 2 (2)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (4) | 9 (9) | 1 (2) | 6 (7) | 8 (10) | 3 (4) | 3 (3)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implant site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 2 (3)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum sickness-like reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chemical eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (5)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 8 (9) | 0 (0) | 5 (6) | 4 (4) | 3 (5) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 5 (7) | 1 (2) | 5 (9)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 5 (6) | 0 (0) | 1 (1)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1) | 3 (5) | 3 (3) | 0 (0) | 1 (2)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (9) | 2 (2) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated for business reasons and not due to any safety or efficacy concerns related to dalotuzumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation and can delete information identified as confidential prior to submission.